CLINICAL TRIAL: NCT02726594
Title: Evaluation of Patient Comfort and Image Quality in Magnetic Resonance Imaging
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Gustav Andreisek, PD Dr. med., University of Zurich
Other Study IDs: KEK-ZH-Nr. 2015-0081
Record Dates: First submitted 2016-03-29; First posted 2016-04-01 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: Patient Satisfaction, Diagnostic Accuracy
Keywords: Magnetic Resonance Imaging, Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients: For the present study, patients who are assigned to the clinically indicated MRI scan, as well as healthy subjects will be included. Healthy volunteers will be recruited through public notices (flyer) (mainly in the district of the University Zurich / USZ). For all patients, the duration of clinical MRI routine examination is 30-90 minutes, depending on the requirements to answer the clinical question. The subjects are interviewed after the MRI scan by a visual analog scale oral and written on various aspects of their perception during the examination. This means an additional expenditure of time of about 10 minutes. The patients arises except for this additional time not a disadvantage by taking part in the study.
- Subjects: For the present study, patients who are assigned to the clinically indicated MRI scan, as well as healthy subjects will be included. Healthy volunteers will be recruited through public notices (flyer) (mainly in the district ETH / USZ). For all patients, the duration of clinical MRI routine examination is 30-90 minutes, depending on the requirements to answer the clinical question. The subjects are interviewed after the MRI scan by a visual analog scale oral and written on various aspects of their perception during the examination. This means an additional expenditure of time of about 10 minutes. The patients arises except for this additional time not a disadvantage by taking part in the study.

SUMMARY:
The aim of this prospective monocentric study is to evaluate the patient comfort in MRI and to measure examination conditions and factors that may affect the image quality and thus the diagnostic accuracy. For this purpose a total of 1000 participants enrolled in the study, consisting of healthy volunteers (N = 300) as well as patients (N = 700), that are assigned to the clinically indicated MRI scan. In this study, individual regions of the body are studied by MRI (for example, knee, ankle, head or spine). For all participants of the study, the investigation for each region examined is exactly the same except that a single external factor is changed or is different. Such variable factors may include: the tube diameter of the magnet, weight of the coil, which is closely attached to the examined area of the body, the height adjustment of the table on which the participants lie, the duration of the study protocol and the generated volume during the investigation. Participants are involuntarily subjected to the particular MRI scanner and setting by availability of USZ Radiology disposition. For the evaluation of the data, participants will be matched in terms of the body regions being examined and based on being part of the patient or subject group. Due to the fine different experimental conditions, the influence of these factors on study patient comfort, as wells as the image quality and thus the diagnostic accuracy will investigated. By this approach, the relevant factors will be examined in isolation. Only by exploring the patient's perception/comfort during an MRI scan, the patient-orientated design of the study conditions can be improved and thus the possibilities of modern MRI technology can be fully utilized in clinical practice.

DETAILED DESCRIPTION:
Background: Magnetic resonance imaging ( "MRI") is an integral part of medical diagnostics since 20 years. Using MRI soft tissue imaging of body regions such as the brain, abdominal or musculoskeletal, is possible and is clearly superior to other imaging techniques. Due to the complex physical conditions a typical MRI scan will take 30-90 minutes (during which the patient should not do any movements), generates a noise level of 75-100 decibels and requires the placement of the patient in an often as cramped perceived tube scanner. These adverse conditions are not only known to have a significantly negative impact on the patient's comfort, but can also change the image quality and thus reduce the diagnostic accuracy of an investigation.

Motivation: At the University Hospital Zurich (USZ) a total of 10, partly very different MR scanners, are available for clinical imaging. These devices differ by the manufacturer and by the different design of the premises, the equipment, the coil and the table sizes, the logs up to the generated in the examination volume and the room temperature. For example, one of the existing examination rooms at the USZ has been equipped by a manufacturer with a costly patient comfort package. This room serves as a showroom and as a positive example for maximum patient comfort. Our experience shows that, overall, all the MRI scans of all units and the resulting image quality fluctuates greatly and the Patient Feedback for the individual studies is partly quite negative. Improved study conditions are therefore accessible both in terms of patient comfort and improved diagnostic accuracy, our goal.

Current status of research: The working group "Research in Musculoskeletal Radiology" at the Institute for Diagnostic and Interventional Radiology at the University Hospital Zurich is led by PhD Dr. med. Gustav Andreisek and under his authority already carried out successfully numerous projects in the field of magnetic resonance imaging.

Objectives: The aim of this prospective monocentric study is to evaluate the patient comfort in MRI and to measure examination conditions and factors that may affect the image quality and thus the diagnostic accuracy. For this purpose a total of 1000 participants enrolled in the study, consisting of healthy volunteers (N = 300) as well as patients (N = 700), which are assigned to the clinically indicated MRI scan. In this study, individual regions of the body are studied by MRI (for example, knee, ankle, head or spine). For all participants in the study, the investigation for each region examined is exactly the same except that a single external factor is changed or is different. Such variable factors may include: the tube diameter of the magnet, weight of the coil, which is closely attached to the examined area of the body, the height adjustment of the table on which the participants lie, the duration of the study protocol and the generated volume during the investigation. Participants are involuntarily subjected to the particular MRI scanner and setting by availability of USZ Radiology disposition. For the evaluation of the data, participants will be matched in terms of the body regions being examined and based on being part of the patient or subject group. Due to the fine different experimental conditions, the influence of these factors on study patient comfort, as wells as the image quality and thus the diagnostic accuracy will investigated. By this approach, the relevant factors will be examined in isolation. Only by exploring the patient's perception/comfort during an MRI scan, the patient-orientated design of the study conditions can be improved and thus the possibilities of modern MRI technology can be fully utilized in clinical practice.

ELIGIBILITY:
Inclusion criteria:

* acceptance of study participation
* age ≥ 18 years.

Exclusion criteria:

* General established contraindications for MRI (i.e. pacemaker implantation with non-compatible pacemakers and pacemaker leads, implantation of other non-MRI-compatible medical devices, metal parts in the body, etc.)
* A pregnancy constitutes an exclusion criterion. If there could be a potentially pregnancy, a pregnancy test will be performed
* claustrophobia

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Overall, 1,000 participants will be included in the study, consisting of healthy volunteers (N = 300) as well as patients (N = 700).
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-08; Primary Completion 2018-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Patient comfort | procedure
  by questionnaires

SECONDARY OUTCOMES:
Image quality | procedure
  by analysis of MRI images

CONTACTS AND LOCATIONS:
Overall Officials: Gustav Andreisek, PD Dr. med., Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No